CLINICAL TRIAL: NCT04179071
Title: An Open-Label, Randomised, Two Part, Two Treatment Crossover Study in Healthy Subjects to Assess the Pharmacokinetics of Savolitinib When Administered Alone and in Combination With Famotidine
Brief Title: A Study in Healthy Male Subjects to Understand How Savolitinib Behaves Inside the Body (Pharmacokinetics) When Administered Alone and in Combination With Famotidine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D5084C00005
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Solid Tumours
Keywords: Famotidine; Drug-drug interaction study; Small molecule kinase inhibitor
MeSH Terms: interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Savolitinib (Experimental): Subjects will receive single dose of 600mg savolitinib after a high-fat, high-calorie meal.
  Interventions: Drug: Savolitinib
- Savolitinib + Famotidine (Experimental): Subjects will receive savolitinib 600mg single dose after high-fat, high-calorie meal and after 1.5 hours (Part A) or 5.5 hours (Part B) of famotidine 40mg dose. Famotidine will be administered after an overnight fast of at least 8 hours with approximately 240 mL of water.
  Interventions: Drug: Savolitinib; Drug: Famotidine

INTERVENTIONS:
Drug: Savolitinib — Subject will receive savolitinib tablet 600mg orally after a high-fat, high-calorie meal.
Drug: Famotidine — Subjects will receive famotidine tablet 40mg orally after an overnight (minimum 8hours) of fasting.
  Arms: Savolitinib + Famotidine

SUMMARY:
This will be an open-label, randomised, 2 part (Part A and Part B), 2 treatment (savolitinib alone or in combination with famotidine), crossover study in healthy, non Japanese, male subjects, performed at a single study centre.

DETAILED DESCRIPTION:
Parts A and B will each have 2 Periods (Period 1 and Period 2) with a crossover design. Part B will be conducted only if results of Part A suggest a clinically meaningful effect of famotidine on savolitinib pharmacokinetics (PK) parameters. In both parts subjects will be randomly assigned 1:1 to receive one of the 2 treatment sequences: savolitinib alone first followed by crossover to the combination treatment of savolitinib+famotidine, or the reverse sequence. Subjects will be admitted for 4 days from one day before the first dose of the study drug and discharged 2 days after. There will be a washout period (no study treatment) of 14 days between the 2 Periods. The essential difference between the 2 parts is that in the combination treatment, famotidine will be administered 2 hours before savolitinib in Part A and 6 hours before savolitinib in Part B. A given subject will receive a total of 1 dose of famotidine and 2 doses of savolitinib during the study.

In this 2 part study, 16 subjects will be randomised in each part to ensure at least 14 evaluable subjects at the end of the last study period. If Part B is conducted, a total of 32 subjects overall are planned to be enrolled in the study. Additional subjects may be enrolled to ensure 14 evaluable subjects in each part if more than 2 subjects are deemed non evaluable.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated written informed consent prior to any study specific procedures.
* Healthy, non-Japanese male subjects with suitable veins for cannulation or repeated venipuncture: male subjects aged 18 to 65 years (inclusive).
* Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive; and weigh at least 50 kg and no more than 100 kg inclusive.
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and total bilirubin (TBL) less than or equal to the upper limit of normal for the institution.
* Have a calculated creatinine clearance greater than 80 mL/min using the Cockcroft-Gault formula at screening.
* Provision of signed, written and dated informed consent for optional genetic/biomarker research. If a subject declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this protocol.

Exclusion Criteria:

* Subject that has at least 1 parent or grandparent (maternal or paternal) of Japanese ethnicity.
* Subjects who screen positive for Helicobacter pylori bacteria.
* History of any clinically significant disease or disorder which, in the opinion of the Principal Investigator (PI), may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of either study drug (savolitinib or famotidine).
* Planned in-patient surgery, dental procedure, or hospitalisation during the study.
* Any clinically important abnormalities in clinical chemistry, haematology, or urinalysis results, as judged by the PI.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
* Abnormal vital signs, after 5 minutes supine rest, defined as any of the following:

  1. Systolic BP <90 mmHg or ≥140 mmHg
  2. Diastolic BP <50 mmHg or ≥90 mmHg
  3. Heart rate <45 or >85 beats per minute.
* Any clinically important abnormalities in rhythm, conduction or morphology of the 12 lead resting electrocardiogram (ECG) that may interfere with the interpretation of QTc interval changes. These include healthy subjects with any of the following:

  1. Abnormal ST-T-wave morphology, particularly in the protocol-defined primary lead (V2) or left ventricular hypertrophy.
  2. PR interval shortening <120 ms (PR >110 ms but <120 ms is acceptable if there is no evidence of ventricular pre-excitation).
  3. PR interval prolongation (>200 ms). Intermittent second (Type 1 second degree block [Wenckebach Phenomenon] while asleep is not exclusive]) or third degree atrioventricular (AV) block, or AV dissociation.
  4. Persistent or intermittent complete bundle branch block, incomplete bundle branch block, or intraventricular conduction delay with QRS >110 ms. Subjects with QRS >110 ms but <115 ms are acceptable if there is no evidence of eg, ventricular hypertrophy or pre-excitation.
  5. Mean resting prolonged QTcF >450 ms or shortened QTcF <340 ms obtained from 3 ECGs.
* A history of additional risk factors for torsades de pointes (TdP) (eg, heart failure, chronic hypokalaemia not correctable with supplements, congenital or familial long QT syndrome, or family history of unexplained sudden death under 40 years of age in first-degree relatives).
* Use of any medications known to prolong the QT/QTc interval and cause TdP.
* Use of any prescribed or non prescribed medication including antacids, analgesics (other than ibuprofen up to 72 hours before dosing day), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of either study drug or longer if the medication has a long half life.
* Known or suspected history of drug abuse, as judged by the PI.
* Current smokers or those who have smoked or used nicotine products within the previous 30 days.
* History of alcohol abuse or excessive intake of alcohol as judged by the PI.
* Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) as judged by the PI.
* Use of drugs with enzyme inducing properties such as St John's Wort, within 3 weeks prior to the first administration of either study drug.
* Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first admission on Day -1.
* Positive screen for drugs of abuse or cotinine (nicotine) or alcohol at screening and before each admission to the Study Centre.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI, or history of hypersensitivity to drugs with a similar chemical structure or class to savolitinib or famotidine.
* Plasma donation within 1 month of screening or any blood donation or loss of >500 mL during the 3 months prior to screening.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of either study drug in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest. Note: subjects consented and screened, but not randomised in this study or a previous Phase I study, are not excluded.
* Subjects who have previously received savolitinib.
* Involvement of any AstraZeneca, Parexel, or study site employee or their close relatives.
* Judgment by the PI that the subject should not participate in the study if they have any ongoing or recent (ie, during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Subjects who are vegans or vegetarians, or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the PI.
* Vulnerable subjects, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* In addition, any of the following is regarded as a criterion for exclusion from the genetic research:
* In addition, the following are considered criteria for exclusion from the optional genetic component of the study:
* Previous bone marrow transplant.
* Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection or previous bone marrow transplant.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) ratio | At pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose on Day 1-3 and Day 16-18
  Cmax ratio of test treatment (savolitinib+famotidine) relative to reference treatment (savolitinib alone) to assess effect of the gastric acid modifier, famotidine, on the PK of savolitinib.
Area under plasma concentration-time curve from zero to infinity (AUC) ratio | At pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose on Day 1-3 and Day 16-18
  AUC ratio of test treatment (savolitinib+famotidine) relative to reference treatment (savolitinib alone) to assess effect of the gastric acid modifier, famotidine, on the PK of savolitinib.

SECONDARY OUTCOMES:
Number of subjects with having adverse events and/or abnormal findings in vital signs and/or laboratory evaluation and/or physical examination | From 28-day screening period to follow-up period i.e. 60 days
  To investigate the safety and tolerability of savolitinib in combination with famotidine.
AUC geometric means ratio of test treatment (savolitinib+famotidine) relative to reference treatment (savolitinib alone) | At pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose on Day 1-3 and Day 16-18
  To assess the effect of famotidine on the PK of savolitinib metabolites M2 and M3 and to describe the PK parameters and the PK concentration-time profiles for savolitinib, M2, and M3 when savolitinib is administered alone and in combination with famotidine.
Area under the plasma concentration curve from time zero to time of last quantifiable concentration AUC(0-t) | At pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose on Day 1-3 and Day 16-18
  AUC(0-t) geometric means ratio of test treatment (savolitinib+famotidine) relative to reference treatment (savolitinib alone) to assess the effect of famotidine on the PK of savolitinib metabolites M2 and M3 and to describe the PK parameters and the PK concentration-time profiles for savolitinib, M2, and M3 when savolitinib is administered alone and in combination with famotidine.
Cmax geometric means ratio of test treatment (savolitinib+famotidine) relative to reference treatment (savolitinib alone) | At pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose on Day 1-3 and Day 16-18
  To assess the effect of famotidine on the PK of savolitinib metabolites M2 and M3 and to describe the PK parameters and the PK concentration-time profiles for savolitinib, M2, and M3 when savolitinib is administered alone and in combination with famotidine.
Cmax metabolite-to-parent ratios (MRCmax) | At pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose on Day 1-3 and Day 16-18
  MRCmax ratio of test treatment (savolitinib+famotidine) relative to reference treatment (savolitinib alone) to assess the effect of famotidine on the PK of savolitinib metabolites M2 and M3 and to describe the PK parameters and the PK concentration-time profiles for savolitinib, M2, and M3 when savolitinib is administered alone and in combination with famotidine.
AUC metabolite-to-parent ratios (MRAUC) | At pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose on Day 1-3 and Day 16-18
  MRAUC ratio of test treatment (savolitinib+famotidine) relative to reference treatment (savolitinib alone) to assess the effect of famotidine on the PK of savolitinib metabolites M2 and M3 and to describe the PK parameters and the PK concentration-time profiles for savolitinib, M2, and M3 when savolitinib is administered alone and in combination with famotidine.
AUC(0-t) metabolite-to-parent ratios [MRAUC(0-t)] | At pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose on Day 1-3 and Day 16-18
  MRAUC(0-t) ratio of test treatment (savolitinib+famotidine) relative to reference treatment (savolitinib alone) to assess the effect of famotidine on the PK of savolitinib metabolites M2 and M3 and to describe the PK parameters and the PK concentration-time profiles for savolitinib, M2, and M3 when savolitinib is administered alone and in combination with famotidine.
Time to reach maximum observed plasma concentration (tmax) | At pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose on Day 1-3 and Day 16-18
  tmax ratio of test treatment (savolitinib+famotidine) relative to reference treatment (savolitinib alone) to assess the effect of famotidine on the PK of savolitinib metabolites M2 and M3 and to describe the PK parameters and the PK concentration-time profiles for savolitinib, M2, and M3 when savolitinib is administered alone and in combination with famotidine.
Half-life associated with terminal slope (λz) of a semi logarithmic concentration-time curve (t½,λz) | At pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose on Day 1-3 and Day 16-18
  t½,λz ratio of test treatment (savolitinib+famotidine) relative to reference treatment (savolitinib alone) to assess the effect of famotidine on the PK of savolitinib metabolites M2 and M3 and to describe the PK parameters and the PK concentration-time profiles for savolitinib, M2, and M3 when savolitinib is administered alone and in combination with famotidine.
Terminal elimination rate constant (λz) | At pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose on Day 1-3 and Day 16-18
  λz ratio of test treatment (savolitinib+famotidine) relative to reference treatment (savolitinib alone) to assess the effect of famotidine on the PK of savolitinib metabolites M2 and M3 and to describe the PK parameters and the PK concentration-time profiles for savolitinib, M2, and M3 when savolitinib is administered alone and in combination with famotidine.
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | At pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose on Day 1-3 and Day 16-18
  Vz/F ratio of test treatment (savolitinib+famotidine) relative to reference treatment (savolitinib alone) to assess the effect of famotidine on the PK of savolitinib metabolites M2 and M3 and to describe the PK parameters and the PK concentration-time profiles for savolitinib, M2, and M3 when savolitinib is administered alone and in combination with famotidine.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | At pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, and 48 hours post-dose on Day 1-3 and Day 16-18
  CL/F ratio of test treatment (savolitinib+famotidine) relative to reference treatment (savolitinib alone) to assess the effect of famotidine on the PK of savolitinib metabolites M2 and M3 and to describe the PK parameters and the PK concentration-time profiles for savolitinib, M2, and M3 when savolitinib is administered alone and in combination with famotidine.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ronald Goldwater, MD, Principal Investigator — Parexel Early Phase Clinical Unit Baltimore (Study Centre)
Locations (1):
- Research Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home